CLINICAL TRIAL: NCT00694057
Title: A Phase II, Double Blind, Randomized, Placebo-Controlled Study of the Safety, Tolerance and Activity of HE3286 When Administered Orally for 12 Weeks to Adult Patients With Type 2 Diabetes Mellitus
Brief Title: Safety, Tolerance and Activity of HE3286 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harbor Therapeutics (Industry)
Responsible Party: Dwight Stickney, MD - Chief Medical Officer, Hollis-Eden Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE3286-0401
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Metformin; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 17-ethynyl-5-androstene-3, 7, 17-triol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsules BID
  Interventions: Drug: Placebo
- Active (Experimental): HE3286 10 mg (5 mg BID)
  Interventions: Drug: HE3286

INTERVENTIONS:
Drug: HE3286 — HE3286 10 mg per day (5 mg BID)
  Arms: Active
Drug: Placebo — Placebo capsules BID
  Arms: Placebo

SUMMARY:
This is a phase II, double-blind, randomized, placebo-controlled study of the safety, tolerance and activity of HE3286 in patients with type 2 diabetes mellitus. Patients receiving stable metformin or who are drug-naive will receive study treatment (HE3286 or placebo) for a treatment period of 12-weeks.

DETAILED DESCRIPTION:
Hollis-Eden Pharmaceuticals, Inc. is developing a new class of therapeutics for the treatment of Type 2 diabetes. The investigational drug, HE3286, holds the potential to be the first in a new class of insulin sensitizers with a potentially novel mechanism of action that may improve the current therapeutic options available to a T2DM patient.

This is a phase II, double-blind, randomized, placebo-controlled study of the safety, tolerance and activity of HE3286 in patients with type 2 diabetes mellitus. Patients receiving stable metformin or who are drug-naive will receive study treatment (HE3286 or placebo) for a treatment period of 12-weeks. Changes in hemoglobin A1c (HbA1c) will be assessed over a treatment period of 12-weeks.

ELIGIBILITY:
Main Inclusion Criteria:

* Patient with a diagnosis of Type 2 Diabetes Mellitus (T2DM)
* Patient must be a) on a stable dose of metformin as monotherapy for at least 10 weeks prior to screening; or b) drug-naive, defined as never having received drug treatment for T2DM or not having received antidiabetic drug therapy during the 3 months prior to screening.
* Patient with a fasting blood glucose level of ≤ 225 mg/dL at screening (≤ 255 mg/dl for drug-naive patients);
* Patient with HbA1c levels >7.5% (7.0 - 10.5% for drug-naive patients) at screening;
* Patient with BMI 28-37 kg/m2 for females 28-39 kg/m2 for males

Main Exclusion Criteria:

* Patient who has a history of clinically significant cardiovascular disease (including coronary artery disease), clinically significant hepatic, respiratory or renal abnormalities within 6 months prior to screening;
* Patient with unstable diabetic complications requiring treatment or ongoing active intervention;
* Patient with a history of long term insulin therapy within the past year;
* Patient who has had therapy with rosiglitazone, pioglitazone, exendin-4 or sitagliptin, alone or in combination within 6 months prior to screening;
* Patient who has any clinically significant abnormalities in laboratory results at screening;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the change in HbA1c from baseline to week 12 in the HE3286 treated group when compared to the placebo group. | 12-weeks
To evaluate the safety and tolerance of HE3286 10 mg per day (5 mg BID) compared to placebo from baseline to week 12. | 12-weeks

SECONDARY OUTCOMES:
To evaluate the effect of HE3286 on fasting blood glucose over time. | 12-weeks
To evaluate the effect of HE3286 on insulin sensitivity over time. | 12-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dwight R. Stickney, MD, Study Director — Harbor Therapeutics
Locations (20):
- United States (20):
  - Anaheim, California
  - Beverly Hills, California
  - Buena Park, California
  - Burbank, California
  - Carmichael, California
  - Escondido, California
  - Fresno, California
  - Huntington Park, California
  - Long Beach, California
  - Los Angeles, California
  - National City, California
  - Roseville, California
  - Chicago, Illinois
  - Baton Rouge, Louisiana
  - St Louis, Missouri
  - Las Vegas, Nevada
  - El Paso, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Kenosha, Wisconsin